CLINICAL TRIAL: NCT05038150
Title: Phase I/IIa, Open-label Study to Evaluate Safety, Tolerability and Preliminary Efficacy of Modified Salmonella Typhimurium SGN1 in Patients With Advanced Solid Tumor
Brief Title: Study of SGN1 in Patients With Advanced Solid Tumor
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangzhou Sinogen Pharmaceutical Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN-P01-001
Record Dates: First submitted 2021-08-24; First posted 2021-09-08 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: The study will employ a standard 3 + 3 escalating dose design to explore dose limiting toxicities (DLTs). Currently plans to evaluate 5 cohorts with 3- 6 patients to determine the Maximum Tolerated Dose (MTD). Patients who had no dose-limiting toxicities observed in Part 1 proceeded to Part 2.
  Alternatively, if a DLT occurs in only 1/3 patients at any dose, then 3 more patients should be enrolled at this dose level. If this is the highest dose and there have been no DLTs-then 3 more patients must be evaluated at the same dose level to confirm the MTD. The MTD is defined as the highest dose at which no more than one (1) DLT is observed among 6 patients.
  Part 3 is an open-label, dose expansion phase. There will be at least 2 tumor types selected , expand between second to four dose level in each tumor type.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort (Experimental): In part 1&2, cohorts of 3 patients will be enrolled. The first patient of each cohort in Part 1 will be admitted to an infusion unit and treated with an IV infusion of SGN1 over 2 hours. Patients in Part 1 will enter Part 2 for extension treatment after completing the 28-day DLT observation period. Up to 5 cohorts will be evaluated.
  Part 3 is an open-label, dose expansion phase.There will be at least 2 tumor types selected, expand between second to four dose level in each tumor type .
  Interventions: Drug: SGN1

INTERVENTIONS:
Drug: SGN1 — The study drug, SGN1, will be administered as an IV infusion through a dedicated line catheter over 2 hours, which unit dose strength is 0.9-2.0×109 cfu /vial.
  Other Names: SalMet-Vec

SUMMARY:
Objectives:To assess the safety and tolerability followed by a dose expansion study to characterize safety, and preliminary efficacy of SGN1 in participants with refractory solid tumors.

Study Rationale:The mechanism of action for SGN1 is based on the fact that most tumors are methionine dependent. SGN1 is designed to be used as a tumor therapeutic bacterium that can preferentially replicate and accumulate in tumors and starve them of essential amino acids by delivering the oncolytic enzyme L-Methioninase.

Patient Population:The treatment populations shall be patients presenting with histologically confirmed advanced and/or metastatic solid tumors that are refractory to standard therapy and for which no other conventional therapy exists.

DETAILED DESCRIPTION:
Methionine starvation can powerfully modulate DNA methylation, cell cycle transition, polyamines and antioxidant synthesis of tumor cells, in contrast to normal ones. L-Methioninase is a pyridoxal phosphate dependent enzyme that catalyzes the γ-elimination reaction of L-methionine to methanethiol, α-ketobutyrate and ammonia. Absolute-dependency on exogenous supply of L-methionine, not homocysteine, for growth and proliferation of tumors is the pivotal biochemical criterion for various human cancers.

SGN1 is a genetically modified strain of Salmonella enterica, serotype typhimurium that expresses L-Methioninase. The attenuated live bacterium has been investigated in China for utility in treating advanced solid tumors. The mechanism of action for SGN1 is based on the fact that most tumors are methionine dependent. SGN1 is designed to be used as a tumor therapeutic bacterium that can preferentially replicate and accumulate in tumors and starve them of essential amino acids by delivering the oncolytic enzyme L-Methioninase.

This study is a multi-center phase I/IIa clinical trial with 3 parts:

Part 1 & 2 is an open-label, dose escalation phase. Part 1 is the DLT observation period, and the patients will enter part 2 for extension treatment after completing the DLT observation period.

Part 3 is an open-label, dose expansion phase. In part 2, the treatment may be terminated if the patients withdraws, has unacceptable toxicity, develops disease progression, experiences an AE that cannot be resolved with/without rescue medication and cause stopping study drug for 2 planned administrations, death, or loss to follow-up. In such cases, patients will be discontinued and palliative or rescue therapy will be offered to those that terminate early.

In part 3, there will be at least 2 tumor types selected, expand between second to four dose level in each tumor type.The Part 3 (Dose expansion stage study) could be started according to the SMC evaluation, do not need waiting the completion the whole cohort of dose escalation (Part 1).

ELIGIBILITY:
Inclusion Criteria

Patients must meet all the following inclusion criteria:

1. Age 18-75 years inclusive of end value, regardless of gender.
2. Part 1: Patients with advanced stage (unresectable or metastatic) cancer including but not limited to small cell lung cancer, non-small cell lung cancer (adeno- and squamous), Hodgkin's lymphoma or non-Hodgkin's lymphoma, sarcoma, cervical carcinoma, melanoma, head and neck cancer, breast cancer, ovarian cancer, pseudomyxoma peritoneum (Pseudomyxoma peritonei, PMP) and hepatocellular carcinoma characterized by failure of standard treatment (disease progression or intolerance, such as chemotherapy, targeted therapy, and other immunotherapies) or patients who have no standard treatment or patients who are intolerant to the standard treatment.

   Part 3: The specific tumor-type expansion study may enroll the following patients: Patients with hepatocellular carcinoma, small cell lung cancer (SCLC), non small cell lung cancer (NSCLC), pancreatic cancer, prostate cancer, bladder cancer, nasopharyngeal carcinoma, sarcoma, melanoma or other tumor type with potential efficacy signal observed in Part 1&2, who have failed to standard therapy or who are intolerant to the standard treatment. There will be 2-4 cohorts of dose expansion in specified tumor types.

   Note: For all tumor species included, standard treatment will refer to current CSCO/NCCN guidelines.

   Standard treatment failure refers to patients who have disease progression after CSCO/NCCN guidelines recommended existing standard care, or relapse/metastasis after standard care.

   Nonstandard treatment refers to patients who have received the treatment recommended by the guidelines and currently have no other effective treatment options.
3. Patients finished anti-tumor therapy including chemotherapy, immunotherapy, biological agents, hormone therapy, radiotherapy (except local radiotherapy for pain relief) ≥ 4 weeks prior to the first dose of study drug.
4. At least 1 measurable lesion according to RECIST 1.1 (for solid tumors).
5. Patients have recovered from any toxic reaction to previous medications (≤Grade 1 based on NCI-CTCAE v 5.0, except a. Hair loss; b. Pigmentation; c. The long-term toxicity caused by radiotherapy and cannot be recovered by the investigator's judgment; d. Platinum induced neurotoxicity of grade 2 and below; e. Hemoglobin at 90 ~ 100 g / L (including boundary value)) or stable status assessed by the investigator.
6. Eastern Co-Operative Oncology Group (ECOG) performance status 0 ~ 1 and a life expectancy of at least 3 months.
7. Laboratory tests must meet the following requirements and have not received any blood cell growth factor 14 days before the test (Patients with laboratory values outside of the specified ranges will be permitted to be retested in order to meet the criteria):

   1. absolute count of neutrophils (ANC) ≥1.5×109 /L, platelet ≥75×109 /L; Hemoglobin ≥90 g/L;
   2. serum albumin ≥30g /L; Bilirubin ≤1.5 × Upper Limit of Normal (ULN), ALT and AST ≤2.5 × ULN;
   3. In patients with liver metastasis,ALT and AST≤5 × ULN;
   4. Creatinine clearance ≥50 mL/min (standard Cockcroft -Gault formula) or Cr ≤1.5 ×ULN: urinary protein≤ 2+ or urinary protein quantitative <1.0 g/L;
   5. International standardized ratio of coagulation function (INR) ≤1.5 × ULN, activated partial thromboplastin time (APTT) ≤1.5 × ULN (If patient has concomitant medication with anticoagulants, whether the coagulation function is qualified will be determined by Investigator.)
8. If female, be either postmenopausal for at least 1 year with documented follicle stimulating hormone (FSH) > 30 IU/L, or surgically sterile for at least 3 months, or if a woman of childbearing potential, must be non-pregnant confirmed by blood and urine pregnancy tests, and non-lactating.
9. Female patients of childbearing potential must agree to use acceptable method(s) of contraception from consent through at least 6 months after last dose of drug infusion.
10. Male patients of reproductive capacity must agree to use effective contraception from start of mobilization through at least 6 months after last dose of drug infusion.
11. Patients with chronic HBV infection with active disease who meet the criteria for anti HBV therapy (HBV DNA test is less than 2000 IU/ml) should be on a suppressive antiviral therapy prior to initiation of cancer therapy. Patients with a history of HCV infection should have completed curative antiviral treatment and HCV viral load below the limit of quantification. Patients with HCV Ab positive but HCV RNA negative due to prior treatment or natural resolution are eligible. Patients on concurrent HCV treatment should have HCV below the limit of quantification.
12. Patients must be able to follow up after the treatment.
13. Patients must understand and voluntarily sign the informed consent form.

Exclusion Criteria

Patients will be excluded from participation for any of the following criteria:

1. Received systemic or absorbable dosage of steroid hormone (prednisone or equivalent) of > 10 mg/day in the 14 days prior to enrollment;

   1. Prednisone > 10 mg/day
   2. Dexamethasone > 1.5 mg/day.
2. Allergic or intolerant to salmonella sensitive antibiotics, or combined with infectious diseases and currently using antibiotics.
3. Present assessable tumors in hollow organs (Stomach, esophagus, intestine, urinary tract etc.).
4. Present with symptomatic central nervous system metastasis or brain abscess at screening.
5. Present with diverticulitis or conditions at screening that might promote the unintentional growth of anaerobic bacteria in non target lesions.
6. Existing cardiac clinical symptoms or diseases that cannot be well controlled, such as:

   1. NYHA grade 2 or above heart failure;
   2. Unstable angina pectoris;
   3. Myocardial infarction occurred within 1 year;
   4. Patients with supraventricular or ventricular arrhythmias that have clinical significance and need treatment or intervention;
   5. Uncontrolled hypertension (systolic blood pressure) ≥160 mmHg and (diastolic blood pressure) ≥100 mmHg after drug treatment;
   6. Patients with valvular heart disease or mitral valve prolapse, aortic valve disease or other source of turbulent cardiac blood flow.
7. Those who had received radiotherapy, chemotherapy, hormone therapy, surgery or molecular targeted therapy that ended fewer than 4 weeks before the first dose of study treatment (if nitrosourea or mitomycin chemotherapy, the interval between end of chemotherapy and first dose of study treatment must be no less than 6 weeks).
8. Patients with active or uncontrolled infection or fever, > 38.5℃, of unknown cause during screening or before the first administration of the study drug (according to the judgment of the researcher, fever caused by tumor can be included).
9. Positive for the presence of human immunodeficiency virus-1 (HIV-1) or human immunodeficiency virus-2 (HIV-2) (positive antigen/antibody and nucleic acid tests); or follow standard of care for HIV diagnosis.
10. Patients with Anti-TP positive.
11. Patients participating in other clinical studies or participating in other clinical studies within 4 weeks (or 5 half-lives of other study drugs), whichever is longer, prior to enrollment and receiving experimental drug administration.
12. Vaccination within 28 days of the first trial treatment, except for administration of inactivated vaccines and RNA vaccines (e.g., inactivated influenza vaccines and COVID-19 RNA vaccines).
13. Received live or attenuated vaccines within 4 weeks of study drug administration, during treatment, or within 5 months of the last administration.
14. In the judgment of the investigator, there are other factors that may lead to termination: for example, adrenal cortex insufficiency, pituitary insufficiency after treatment, and other serious diseases (including 14.mental diseases) need to be treated together, there are serious abnormalities in laboratory examination, family or social factors, which may affect the safety of the patients or test data and sample collection.
15. In the researcher's judgment, patients who are not suitable for other reasons.
16. Documented salmonella infections within 6 months.
17. Abdominal standing position plain film or abdominal CT indicates the possibility of bowel obstruction within 6 months from screening, or the Investigator believes there is a risk of bowel obstruction.
18. Patients with implants such as pacemakers, prosthetic cardiac valves, or metal orthopedic prostheses (not include vascular implants for Part 3).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2028-01-18 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of AEs (adverse events). | From receiving study drug and throughout the study, until 28 days after the last dosing.
  An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product and does not imply any judgment about causality.
  Events meeting the definition of an AE include:
  * Any abnormal laboratory test results (hematology, serum chemistry, or urinalysis) or other safety assessments (e.g., ECGs, vital signs measurements), including those that worsen from baseline, and was felt to be clinically significant in the medical and scientific judgment of the Investigator.
  * Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition.
  * New conditions detected or diagnosed after study treatment administration even though it may have been present prior to the start of the study.
  * Signs, symptoms, or the clinical sequelae of a suspected interaction.
Incidence of SAEs. | From receiving study drug and throughout the study, until 28 days after the last dosing.
  An AE or suspected adverse reaction is considered "serious" if it results in any of the following outcomes:
  * Death
  * Life-threatening
  * Inpatient hospitalization or prolongation of existing hospitalization
  * A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  * A congenital anomaly/birth defect
  * Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.
Objective response rate (ORR) | From signing the informed consent form until 28 days after the last dose.
  The efficacy endpoints include ORR, DCR and PFS. The ORR is defined as the proportion of patients who achieve PR or better according to the RECIST v1.1 and Choi, mRECIST is used to assess Hepatocellular carcinoma, and LYRIC is used to assess Lymphoma. as assessed by investigator.
Disease control rate (DCR) | From signing the informed consent form until 28 days after the last dose.
  The efficacy endpoints include ORR, DCR and PFS. The DCR is defined as the proportion of patients who achieve SD or better according to the RECIST v1.1 and Choi , mRECIST is used to assess Hepatocellular carcinoma, and LYRIC is used to assess Lymphoma. as assessed by investigator.
Progress Free Survival (PFS) | From signing the informed consent form until 28 days after the last dose.
  The efficacy endpoints include ORR, DCR and PFS. PFS is defined as the time interval from date of first dose of SGN1 to the date of documented disease progression (iRECIST is used when the subject is suspected to have pseudo disease progression) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Incidence with any dose limiting toxicity (DLT),to determine the MTD. | Up to 28 days post first dose.
  Any of the following judged to be associated with SGN1 (i.e., possibly-, probably-, or definitely related to), may be considered a DLT:
  1. Any Grade 5 adverse event that is at least possibly related to investigational drug.
  2. Non-hematological toxicities:
     1. Grade 4 non-hematological toxicities (excluding alopecia) lasting > 3 days despite optimal supportive care (OSC).
     2. Grade 3 non-hematologic toxicities lasting > 7 days despite optimal supportive care (OSC).
  3. Hematological toxicities:
     1. Grade 4 hematologic toxicity lasting > 7 days (except following b and c).
     2. Grade 3 or 4 febrile neutropenia (body temperature ≥38.5°C) lasting > 7 days.
     3. Grade 3 thrombocytopenia with bleeding or Grade 4 thrombocytopenia.
Incidence with adverse events and preliminary efficacy data to determine the OBD. | From receiving study drug and throughout the study, until 28 days after the last dosing.
  OBD will be determined by adverse events, preliminary efficacy data,and the OBD determined by the SMC.
PK analysis of SGN1 level in blood. | For the first four infusions in Part 1 and Part 3
  Concentrations of SGN1 will be measured. In Part 1 and Part 3, blood sampling for pharmacokinetics analyses will be conducted. The blood collection times for PK are within 30 minutes Pre-dose and immediately end of injection of first 4 infusions (C1D1, C1D8, C1D15 and C1D22);for first and fourth infusion(C1D1 and C1D22) extra blood sample needs to be collected at the following timepoints after the end of infusion procedure: 15 minutes (± 3 minute), 30 minutes (± 3 minute), 45 minutes (± 3 minute), 1 hour (± 5 minutes), 1.5 hours (± 5 minutes), 2 hours (± 5 minutes), 4 hours (± 10 minutes) and every 30 minutes (± 3 minute) during the infusion procedure, besides, after the start time of infusion, following PK timepoints:24 hours ± 1 hour, 48 hours ± 1 hour and 72 hours ± 1 hour for C1D1 and C1D22.PK blood sampling points may be modified based on patients' PK parameters in future.
Bacterial shedding of SGN1 level in blood. | Before the first administration up to 28 days after the last dosing.
  In Part 1 and Part 3 ,SGN1 blood concentrations before and after the first SGN1 infusion are measured in the PK Analysis described above. The qPCR results from PK blood samples will contribute to the analysis as the bacterial shedding of SGN1 in blood.
  For subsequent SGN1 infusions (starting with Dose 2),blood samples shall be collected within 2 hours prior to the start of SGN1 infusion and 24 hours±3 hours post end of infusion.
  If blood samples test positive for SGN1, collection of shedding samples should continue with weekly SGN1 administration until the samples from three consecutive infusions result below the limit of detection (LOD). If samples collected around the first three doses result at or below the limit of detection (LOD), subsequent sample collection and testing is not required.
  In EOT/ET visit, blood samples for bacterial shedding will be collected.
Bacterial shedding of SGN1 level in urine. | Before the first administration up to 28 days after the last dosing.
  In Part 1 and Part 3, for the first SGN1 administration (C1D1), urine sampling for bacterial shedding will be conducted within 2 hours before administration, 3 hours ±1 hour, 6 hours ±1 hour, 24 hours ±3 hours, 48 hours ±3 hours and 72 hours ±3 hours after end of infusion.
  For subsequent SGN1 infusions (starting with Dose 2), urine samples shall be collected within 2 hours prior to the start of SGN1 infusion and within 24 hours ±3 hours post end of infusion.
  If urine samples test positive for SGN1, collection of shedding samples should continue with weekly SGN1 administration until the samples from three consecutive infusions result below the limit of detection (LOD). If samples collected around the first three doses result at or below the limit of detection (LOD), subsequent sample collection and testing is not required.
  In EOT/ET visit, urine samples for bacterial shedding will be collected.
Bacterial shedding of SGN1 level in saliva. | Before the first administration up to 28 days after the last dosing.
  For the first SGN1 administration (C1D1), saliva sampling for bacterial shedding will be conducted within 2 hours before administration, 3 hours ±1 hour, 6 hours ±1 hour, 24 hours ±3 hours, 48 hours ±3 hours and 72 hours ±3 hours after end of infusion.
  For subsequent SGN1 infusions (starting with Dose 2), saliva samples shall be collected within 2 hours prior to the start of SGN1 infusion and within 24 hours ±3 hours post end of infusion. If saliva samples test positive for SGN1, collection of shedding samples should continue with weekly SGN1 administration until the samples from three consecutive infusions result below the limit of detection (LOD). If samples collected around the first three doses result at or below the limit of detection (LOD), subsequent sample collection and testing is not required.
  In EOT/ET visit, saliva samples for bacterial shedding will be collected.
Bacterial shedding of SGN1 level in feces. | Before the first administration up to 28 days after the last dosing.
  Feces samples for bacterial shedding will be collected by the patient before first administration of SGN1; this sample may be collected at any time during the screening period. Additional feces samples are to be collected after the end of the first infusion within the time frames below.
  0-24 hours 24-48 hours 48-72 hours For subsequent SGN1 infusions (starting with Dose 2), will be collected by the subject within 72 hours prior to infusion and within 72 hours after the end of infusion.
  If feces samples test positive for SGN1, collection of shedding samples should continue with weekly SGN1 administration until the samples from three consecutive infusions result below the limit of detection (LOD).If samples collected around the first three doses result at or below the limit of detection (LOD), subsequent sample collection and testing is not required.
  In EOT/ET visit, feces samples will be collected by the subject within 24 hours prior to the EOT/ET visit.
Anti-Drug antibody (ADA) of SGN1. | Before the first administration up to 28 days after the last dosing.
  Collecting of anti-drug antibodies (ADA) blood samples from all patients.
  Blood samples will be collected before the each administration (within 2 days) for first 2 cycles and first administration of 3rd cycle (C1D1~C3D1) and 24 hours (± 6 hours) post infusion for cycle 1 and cycle 2 (C1D2~C2D23), and at the end of treatment/withdrawal visit.
  The Subsequent ADA blood samples collection timepoints will be adjusted according to the subject's ADA analysis result.
Assessment of tumor colonization. | From receiving study drug and throughout the study, until 28 days after the last dosing.
  For appropriate superficial tumors, colonization of the tumor by SGN1 will be assessed by fine needle aspiration and/or excise biopsies every 8 weeks.
Proinflammatory cytokines | Within 7 days prior to the first dose, and at 2, 4, 6, and 24 hours post end of first infusion.
  Proinflammatory cytokines including IL-1β, IFN-γ,TNF-α, IL-6, and IL-8.

OTHER OUTCOMES:
Tumor biomarkers upon cancer types | From baseline until 28 days after the last dose.
  The changes before and after treatment of tumor biomarkers upon cancer types.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (4):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Health Chao Family Comprehensive Cancer Center, Orange, California
  - Barbara Ann Karmanos Cancer Hospital dba Karmanos Cancer Center, Detroit, Michigan
  - University of Cincinnati Cancer Center, Cincinnati, Ohio
- China (4):
  - Guangdong Clifford Hospital, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Shanghai Jiao Tong University Affiliated Sixth People's Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No